CLINICAL TRIAL: NCT03327012
Title: Efficacy and Safety of Panlongqi Tablet in Patients With Knee Osteoarthritis:A Multicenter, Randomized, Double-blind, Placebo-controlled Parallel Study
Brief Title: Efficacy and Safety of Panlongqi Tablet in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director，Devision of Rheumatology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLQ_2016001
Record Dates: First submitted 2017-10-22; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of Panlongqi Tablet (Experimental): Patients were treated with Panlongqi Tablet.
  Interventions: Drug: Treatment of Panlongqi Tablet
- Treatment of Panlongqi Placebo (Placebo Comparator): Patients were treated with Panlongqi Placebo Tablet.
  Interventions: Drug: Treatment of Panlongqi placebo

INTERVENTIONS:
Drug: Treatment of Panlongqi Tablet — Panlongqi Tablet:1.2g,3times a day, oral, for 4 weeks.
  Other Names: capsule A
  Arms: Treatment of Panlongqi Tablet
Drug: Treatment of Panlongqi placebo — Panlongqi placebo:1.2g,3times a day, oral, for 4 weeks.
  Other Names: capsule B
  Arms: Treatment of Panlongqi Placebo

SUMMARY:
This study evaluates the efficacy and safety of Panlongqi tablet compared with placebo in the treatment of knee osteoarthritis in adults.Half of participants will receive Panlongqi tablet in combination,while the other half will receive a Placebo.

DETAILED DESCRIPTION:
The test group will be given Panlongqi tablet 1.2g three times per day,the control group will be given placebo 1.2g three times per day. The invention will last 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1.40-75 years of age (including 40 years and 75 years old), men and women are not limited.

2. western medicine diagnosis of knee osteoarthritis, clinical classification for primary.

3.The severity of the imaging classification of K-L≤Ⅲ; 4. treatment VAS pain scores than 40mm (select the subjects most obvious limb pain symptoms).

5. informed consent form signed by the patient or legal representative.

Exclusion Criteria:

1. within 3 months prior to the trial, the patients were treated within 1 years.
2. 4 weeks before the treatment, corticosteroids, non steroidal drugs, intra-articular injections or other drugs to improve the condition (such as cartilage protective agents) were used.
3. Swelling of the knee joint.
4. knee synovial crystalline (joint) inflammation, acute inflammatory arthritis, rheumatoid arthritis, metabolic bone disease, psoriatic arthritis, septic arthritis, systemic lupus erythematosus, Sjogren syndrome, vasculitis and other rheumatic diseases caused by inflammatory arthritis and endocrine diseases caused by.
5. the screening period has any disease history or evidence: The basic of serious cardiovascular and cerebrovascular diseases; An active, recurrent peptic ulcer or other hemorrhagic disease risk; Sales and other serious diseases of digestive system; An associated with malignant tumors, blood, or other serious diseases or system;
6. patients who are unable to cooperate or cooperate with other mental disorders.
7. before the screening, any laboratory test indicators meet the following standards: An admission of liver and kidney function showed that ALT and AST is more than 1.5 times the upper limit of the normal value, Cr is more than 1.2 times the upper limit of normal (Reference Research Center laboratory where the range of normal value); An other clinically significant laboratory abnormalities, and the researchers judged not into the group.
8. allergic constitution or allergic to test seven tablets, excipients or similar ingredients;
9. doubt or indeed history of alcohol and drug abuse;
10. pregnant or lactating women or recent planned pregnancies and those who are reluctant to use contraceptives;
11. participants who participated in other clinical trials within the first 3 months.
12. the researchers believe that patients should not participate in this clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-03-28 (Estimated); Study Completion 2019-07-28 (Estimated)

PRIMARY OUTCOMES:
The change from Baseline to week 4 in Visual Analog Scale (VAS)score | 0 weeks,2 weeks，4 weeks
  VAS scores ranges from 0 to 100, with higher scores indicating heavier pain

SECONDARY OUTCOMES:
The change from Baseline to week 4 in Western Ontarioand McMaster Universities Osteoarthritis Index (WOMAC)score | 0 weeks,2 weeks and 4 weeks
  WOMAC scores ranges from 0 to 96, with higher scores indicating greater disability
The change from baseline to week 4 in The Short Form-36 Health Survey (SF-36) scores | 0 weeks,4 weeks
  SF-36 scores ranges from 0 to 100,it shows the extent of physical function restriction with higher scores indicating greater disability
The number of adverse events | 4 weeks
  The number of adverse events related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, Doctor, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sc
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided